CLINICAL TRIAL: NCT07194980
Title: Safety and Efficacy of the Addition of Nemtabrutinib to Lisocabtagene Maraleucel in Patients With Relapsed/Refractory Chronic Lymphocytic Leukemia
Brief Title: Nemtabrutinib and Lisocabtagene Maraleucel for the Treatment of Relapsed/Refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1125624; NCI-2025-06406 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20853 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2025-09-19; First posted 2025-09-26 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ARQ531

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (nemtabrutinib, lisocabtagene maraleucel) (Experimental): Patients receive nemtabrutinib PO daily on days 1-28 of each cycle (NOTE: nemtabrutinib is not given during lymphodepleting therapy). Cycles repeat every 28 days for up to 1 year after lisocabtagene maraleucel infusion in the absence of disease progression or unacceptable toxicity. Patients undergo leukapheresis 7 days after start of nemtabrutinib treatment. Patients receive SOC lymphodepleting therapy consisting of cyclophosphamide IV and fludarabine IV on approximately the 5th, 4th, and 3rd day prior to lisocabtagene maraleucel infusion. Patients then receive lisocabtagene maraleucel IV 36-96 hours after completion of SOC lymphodepleting therapy. Patients also undergo TTE or MUGA during screening, and PET/CT scans, bone marrow biopsy and aspiration, lymph node biopsy, and blood sample collection throughout the study.
  Interventions: Drug: Nemtabrutinib; Biological: Lisocabtagene Maraleucel

INTERVENTIONS:
Drug: Nemtabrutinib — Given PO
  Other Names: ARQ 531; ARQ-531; ARQ531; Bruton's Tyrosine Kinase Inhibitor ARQ 531; BTK Inhibitor ARQ 531; MK-1026
Biological: Lisocabtagene Maraleucel — Given IV
  Other Names: Anti-CD19-CAR Genetically Engineered Autologous T Lymphocytes JCAR017; Anti-CD19-CAR Genetically Engineered Autologous T-lymphocytes JCAR017; Autologous Anti-CD19-EGFRt-4-1BB-zeta-modified CAR CD8+ and CD4+ T-lymphocytes JCAR017; Breyanzi; JCAR 017; JCAR-017; JCAR017; Liso-cel

SUMMARY:
This phase II trial studies how well the addition of nemtabrutinib to lisocabtagene maraleucel in treating patients with chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL) that has come back after a period of improvement (relapsed) or that does not respond to treatment (refractory). Nemtabrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Lisocabtagene maraleucel is a type of treatment called chimeric antigen receptor (CAR) T-cell therapy, in which a patient's T-cells (a type of immune system cell) are changed in the laboratory so they will attack cancer cells. T-cells are taken from a patient's blood. Then the gene for a special receptor that binds to a certain protein on the patient's cancer cells is added to the T-cells in the laboratory. The special receptor is called a chimeric antigen receptor (CAR). Large numbers of the CAR T-cells are grown in the laboratory and given to the patient by infusion for treatment. Adding nemtabrutinib to lisocabtagene maraleucel may be an effective treatment for relapsed/refractory CLL/SLL.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive nemtabrutinib orally (PO) daily on days 1-28 of each cycle (NOTE: nemtabrutinib is not given during lymphodepleting therapy). Cycles repeat every 28 days for up to 1 year after lisocabtagene maraleucel infusion in the absence of disease progression or unacceptable toxicity. Patients undergo leukapheresis 7 days after start of nemtabrutinib treatment. Patients receive standard of care (SOC) lymphodepleting therapy consisting of cyclophosphamide intravenously (IV) and fludarabine IV on approximately the 5th, 4th, and 3rd day prior to lisocabtagene maraleucel infusion. Patients then receive lisocabtagene maraleucel IV 36-96 hours after completion of SOC lymphodepleting therapy. Patients also undergo transthoracic echocardiogram (TTE) or multigated acquisition scan (MUGA) during screening, and positron emission tomography (PET)/computed tomography (CT) scans, Bone marrow biopsy and aspiration, lymph node biopsy, and blood sample collection throughout the study.

After completion of study treatment, patients are followed for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CLL/SLL per International Workshop on Chronic Lymphocytic Leukemia (iwCLL) classification
* Measurable disease by imaging (lymph node [LN] > 1.5cm) or absolute lymphocyte count (ALC) (> 5000/μL) or marrow involvement of at least 30% by flow cytometry
* Eligible for lisocabtagene maraleucel (liso-cel) as standard-of-care per Food and Drug Administration (FDA) label for CLL/SLL
* At least 18 years of age at time of study enrollment
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* The ability to swallow and retain oral medication

  * NOTE: Administration of nemtabrutinib is not permitted through a percutaneous endoscopic gastro-jejunal (J PEG) tube
* Participants who are hepatitis B surface antigen (HBsAg) positive are eligible if they have received hepatitis B virus (HBV) antiviral therapy for at least 4 weeks and have undetectable HBV viral load prior to randomization

  * Note: Participants should remain on anti-viral therapy throughout study intervention and follow local guidelines for HBV anti-viral therapy post completion of study intervention. Hepatitis B screening tests should include HBsAg and anti-HBV. Hepatitis B screening tests are not required unless:

    * Known history of HBV infection,
    * As mandated by local health authority
* Absolute neutrophil count (ANC) ≥ 500/µL

  * Growth factor and/or transfusion support is permissible to stabilize participant prior to study treatment if needed
  * No lower limit if cytopenia is related to bone marrow involvement
* Hemoglobin ≥ 8 g/dL

  * Growth factor and/or transfusion support is permissible to stabilize participant prior to study treatment if needed
  * No lower limit if cytopenia is related to bone marrow involvement
* Platelets ≥ 25 000/µL

  * Growth factor and/or transfusion support is permissible to stabilize participant prior to study treatment if needed
  * No lower limit if cytopenia is related to bone marrow involvement
* Creatinine ≤ 1.5 × upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or CrCl) ≥ 30 mL/min for participant with creatinine levels > 1.5 × institutional ULN

  * Creatinine clearance (CrCl) should be calculated per institutional standard
* Total bilirubin ≤ 1.5 × ULN OR direct bilirubin ≤ ULN for participants with total bilirubin levels > 1.5 × ULN
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) ≤ 2.5 × ULN (≤ 5 × ULN for participants with liver metastases)
* International normalized ratio (INR) OR prothrombin time (PT) ≤ 1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants
* Activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Cardiac (echocardiogram [Echo] or multi-gated acquisition scan [MUGA]) ejection fraction ≥ 40%

Exclusion Criteria:

* Diagnosis of Richter Transformation
* Clinically significant (symptomatic) central nervous system (CNS) involvement at time of study enrollment. Previously treated CNS disease is allowed if the participant is asymptomatic. Incidental findings including positive cerebral spinal fluid (CSF) studies are not exclusionary
* Active infection and uncontrolled infection
* Active HBV/hepatitis C virus (HCV) infection

  * Participants must have completed curative anti-viral therapy for HCV at least 4 weeks prior to study enrollment
  * Participants who are HBsAg positive are eligible if they have received HBV antiviral therapy for at least 4 weeks and have undetectable HBV viral load prior to study enrollment
  * Note: Participants should remain on anti-viral therapy throughout study intervention and follow local guidelines for HBV anti-viral therapy post completion of study intervention
* HIV with a detectable viral load or a CD4 count ≤ 350 cells/µL at time of screening

  * Participants with HIV who do not meet the above criteria are eligible if they are on a stable antiretroviral therapy (ART) regimen (ART must not be strong CYP3A4 inducers) for at least 4 weeks prior to study entry and are compliant with ART are eligible
  * Patients with an AIDS defining opportunistic infection in the past 12 months prior to screening
* Gastrointestinal dysfunction that may affect drug absorption (e.g., gastric bypass surgery, gastrectomy)
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator
* Corrected QT interval (QTc) prolongation (defined as a QTc > 450 msecs) or other significant electrocardiogram (ECG) abnormalities including second degree atrioventricular (AV) block type II, third degree AV block, or bradycardia (ventricular rate less than 50 beats/min)
* Known allergy/sensitivity to nemtabrutinib or any of the excipients
* Known prior progressive disease while on nemtabrutinib

  * NOTE: Refer to the investigator's brochure (IB) for details regarding prior recipients of nemtabrutinib
* History of severe bleeding disorder defined as an ongoing congenital or acquired condition that leads to an increased likelihood of bleeding
* History of a second malignancy

  * NOTE: The time requirement does not apply to participants who underwent successful definitive resection of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ, excluding carcinoma in situ of the bladder
* A participant of childbearing potential (POCBP) who has a positive urine pregnancy test within 72 hours prior to study enrollment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required

  * Note: In the event that 72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative in order for participant to start receiving study medication
* Need or anticipation of need for additional bridging therapy in addition to nemtabrutinib

  * Palliative radiation therapy for less than 2 weeks or the use of prednisone 30mg (or the prednisone equivalent) for a maximum of 5 days is allowed and is not exclusionary
* Currently being treated with the following drugs:

  * P-gp substrates with a narrow therapeutic index
  * CYP3A strong inducers
  * CYP3A strong inhibitors
  * NOTE: A washout period of at least 5 times the half-life after the last dose of any of the above treatments is required for a participant to be eligible for study enrollment
* Has received a live vaccine or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of inactivated vaccines are allowed
* Is currently enrolled on another therapeutic clinical trial. Concurrent enrollment on another therapeutic clinical trial or any trial designed to impact the efficacy of anti-cancer therapy is prohibited
* Has received an investigational agent or has used an investigational device within 4 weeks prior to study intervention administration
* Has not adequately recovered after 4 weeks from major surgery or has ongoing surgical complications

  * Note: Biopsy and placement of central venous access devices are not considered major surgery
* Has a history or current evidence of any condition, therapy, or laboratory abnormality or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Any condition or history that the study investigator deems not in the best interest of the patient to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2029-10-20 (Estimated); Study Completion 2029-10-20 (Estimated)

PRIMARY OUTCOMES:
Complete response (CR) | Up to 5 years after completion of study treatment
  Will be defined by the International Workshop on Chronic Lymphocytic Leukemia (iwCLL) criteria. Binary proportions will be estimated along with 95% confidence intervals. Confidence intervals for binary proportions will be estimated using the Wilson Score method.

SECONDARY OUTCOMES:
Overall response rate | Up to 5 years after completion of study treatment
  Will be defined by the iwCLL criteria. Binary proportions will be estimated along with 95% confidence intervals. Confidence intervals for binary proportions will be estimated using the Wilson Score method.
Overall survival (OS) | From first dose of protocol treatment to documentation of the first sign of disease progression or death from any cause, assessed up to 5 years after completion of study treatment
  The distribution of OS will be estimated using the method of Kaplan-Meier. Confidence intervals around median time will be estimated using the Brookmeyer Crowley method.
Progression free survival (PFS) | From first dose of protocol treatment to documentation of the first sign of disease progression or death from any cause, assessed up to 5 years after completion of study treatment
  Will be defined by the iwCLL criteria. The distribution of PFS will be estimated using the method of Kaplan-Meier. Confidence intervals around median time will be estimated using the Brookmeyer Crowley method.
Time to response (TTR) | From start of protocol treatment to first documentation of response among participants documented to have a response, assessed up to 5 years after completion of study treatment
  Will be defined by the iwCLL criteria among responders. The distribution of TTR will be estimated using the method of Kaplan-Meier. Confidence intervals around median time will be estimated using the Brookmeyer Crowley method.
Time to next treatment (TTNT) | From start of protocol treatment to the start of a subsequent treatment, assessed up to 5 years after completion of study treatment
  TTNT is only defined for participants who start a new treatment and only for those participants with progressive CLL/SLL. The distribution of TTNT will be estimated using the method of Kaplan-Meier. Confidence intervals around median time will be estimated using the Brookmeyer Crowley method.
Duration of response (DoR) | From first documentation of response to documentation of the first sign of disease progression or death from any cause, whichever comes first, assessed up to 5 years after completion of study treatment
  Will be defined by the iwCLL criteria among responders. The distribution of DoR will be estimated using the method of Kaplan-Meier. Confidence intervals around median time will be estimated using the Brookmeyer Crowley method.
CR on positron emission tomography/computed tomography by Lugano criteria | Up to 5 years after completion of study treatment
  Binary proportions will be estimated along with 95%. Confidence intervals. Confidence intervals for binary proportions will be estimated using the Wilson Score method.
Incidence of adverse events | Up to 30 days after the last dose of nemtabrutinib
  Will be assessed by Common Terminology Criteria for Adverse Events 5.0.
Incidence of dose-limiting toxicity (DLT) | Up to 28 days following the infusion of lisocabtagene maraleucel
  For the purpose of this study, the initial observed DLT will be considered the event which counts toward safety suspension rules.
Incidence of cytokine release syndrome (CRS) or immune effector cell-associated neurotoxicity (ICANS) | Up to 30 days following the infusion of lisocabtagene maraleucel
  Grade, day of onset, and duration of CRS or ICANS by American Society of Transplant and Cellular Therapy (ASTCT) Consensus grading.
Time to CRS or ICANS onset | Up to 30 days following the infusion of lisocabtagene maraleucel
  Grade, day of onset, and duration of CRS or ICANS by ASTCT Consensus grading. The distribution of time to CRS or ICANS onset will be estimated using the method of Kaplan-Meier. Confidence intervals around median time will be estimated using the Brookmeyer Crowley method.
Time from CRS or ICANS onset to resolution | Up to 30 days following the infusion of lisocabtagene maraleucel
  Grade, day of onset, and duration of CRS or ICANS by ASTCT Consensus grading. The distribution of time from CRS or ICANS onset to resolution will be estimated using the method of Kaplan-Meier. Confidence intervals around median time will be estimated using the Brookmeyer Crowley method.

CONTACTS AND LOCATIONS:
Overall Officials: Mazyar Shadman, MD, MPH, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No